CLINICAL TRIAL: NCT04522349
Title: Randomized Crossover Trial Comparing Shoulder Abduction Movements, Manual Dexterity and Satisfaction of Transradial Amputees Using Axon-Hook and Greifer Myoelectric Hooks.
Brief Title: Compensatory Movements With Axon-Hook and Greifer in Transradial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock France SNC (Industry)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20PT003-FR-01-0516; 2016-A00897-44 (Other: RCB (ANSM))
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Transradial Amputation
Keywords: shoulder compensatory movements; myoelectric hooks; manual dexterity; satisfaction; Axon-Hook; Greifer
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: randomized crossover trial (AB/BA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greifer then Axon-Hook (Active Comparator): T0 + 2 weeks: evaluation with Greifer. T1 + 2 weeks: evaluation with Axon-Hook
  Interventions: Device: Greifer then Axon-Hook
- Axon-Hook then Greifer (Active Comparator): T0 + 2 weeks: evaluation with Axon-Hook. T1 + 2 weeks: evaluation with Greifer
  Interventions: Device: Axon-Hook then Greifer

INTERVENTIONS:
Device: Greifer then Axon-Hook — Each participant is fitted with a Greifer and assessed after two weeks home-trial. Then he is fitted with Axon-Hook and assessed after two weeks home trial.
  Arms: Greifer then Axon-Hook
Device: Axon-Hook then Greifer — Each participant is fitted with a Axon-Hook and assessed after two weeks home-trial. Then he is fitted with Greifer and assessed after two weeks home trial.
  Arms: Axon-Hook then Greifer

SUMMARY:
Upper limb amputees often report musculoskeletal pain due to exaggerated shoulder abduction movements. Previous studies on prosthetic hands showed that wrist orientation contributes to reduce shoulder compensatory movements. The hypothesis of this research is that prosthetic hooks may also provide better functional outcomes when offering wrist adjustments and a design that favors a good visualization of the grips. The objective of this study is to compare shoulder abduction, manual dexterity and satisfaction when using Axon-Hook and Greifer myoelectric hooks during repetitive tasks. Shoulder abduction and manual dexterity results are also compared with the sound side.

DETAILED DESCRIPTION:
Depending on patient's expectations, different prosthetic solutions can be offered. If prosthetic hands, being at the same time functional and aesthetic solutions, are widely used, for some professional or leisure activities, myoelectric users will have a better functional response with a non-morphologic terminal device such as a hook.

Axon-hook and Greifer are two myoelectric hooks proposed by Otto Bock HealthCare. Greifer (Myobock system) has two movable strong hooks and a wrist that can be orientated medially or laterally. Axon-Hook (Axon-Bus system) has thin hooks for a good visualization of the grip, one being fixed for more precision, and a flexible wrist that can be orientated and locked in flexion and extension position.

Previous studies on myoelectric hands showed that functionalities of prosthetic components such as type of hand or type of wrist, have an influence on compensatory movements, which can explain musculoskeletal pains. The hypothesis of the study is that Axon-Hook may reduce shoulder abduction and improve patient satisfaction. No significant difference is expected regarding manual dexterity.

This randomized corossover trial compares shoulder abduction, manual dexterity and satisfaction while using Axon-Hook and Greifer. Shoulder abduction and manual dexterity results are also compared with the sound side.

ELIGIBILITY:
Inclusion Criteria:

* persons with trans-radial upper limb amputation
* persons whose amputation is acquired or congenital
* persons who regularily uses a myoelectric prosthesis and who controls it
* persons whose residual limb is stabilized, with a minimum time of six month since amputation
* persons whose profesional activity or life project justify or could justify the use of a myoelectric hook
* persons who gave their written consent to participate to the study

Exclusion Criteria:

* persons under 18 years of age
* pregnant woman
* persons unable to personnaly give their consent
* persons with psychic or linguistic inability to understand instructions for the test
* persons unavailable to comply with the entire study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Average shoulder abduction measure | One minute
  Average measure of shoulder abuction during Box and Blocks manual dexterity test, by motion analysis

SECONDARY OUTCOMES:
Percentage of time spent with shoulder abduction more or equal to 60° | One minute
  Percentage of time spent with shoulder abduction more or equal to 60° during Box and Blocks test
Manual dexterity | One minute
  Score at the Box and Blocks test
User satisfaction | 15 minutes
  Score at the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Amélie TOUILLET, Principal Investigator — Institut Régional de Rééducation et de Réadaptation de Nancy
Locations (1):
- Institut Régional de Rééducation et de Réadaptation, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A.G. Cutti; I. Parel; M. Luchetti; E. Gruppioni; N. Rossi; G. Verni, The Psychosocial and Biomechanical Assessment of Amputees Fitted with Commercial Multi-grip Prosthetic Hands, in: Grasping the Future: Advances in Powered Upper Limb Prosthetics, BOLOGNA, VINCENZO PARENTI CASTELLI & MARCO TRONCOSSI, 2012, pp. 59 - 77
- [Background] Major MJ, Stine RL, Heckathorne CW, Fatone S, Gard SA. Comparison of range-of-motion and variability in upper body movements between transradial prosthesis users and able-bodied controls when executing goal-oriented tasks. J Neuroeng Rehabil. 2014 Sep 6;11:132. doi: 10.1186/1743-0003-11-132. PMID 25192744
- [Background] Carey SL, Dubey RV, Bauer GS, Highsmith MJ. Kinematic comparison of myoelectric and body powered prostheses while performing common activities. Prosthet Orthot Int. 2009 Jun;33(2):179-86. doi: 10.1080/03093640802613229. PMID 19367522
- [Background] Metzger AJ, Dromerick AW, Holley RJ, Lum PS. Characterization of compensatory trunk movements during prosthetic upper limb reaching tasks. Arch Phys Med Rehabil. 2012 Nov;93(11):2029-34. doi: 10.1016/j.apmr.2012.03.011. Epub 2012 Mar 23. PMID 22449551
- [Background] Ostlie K, Franklin RJ, Skjeldal OH, Skrondal A, Magnus P. Musculoskeletal pain and overuse syndromes in adult acquired major upper-limb amputees. Arch Phys Med Rehabil. 2011 Dec;92(12):1967-1973.e1. doi: 10.1016/j.apmr.2011.06.026. PMID 22133243
- [Background] Bertels T, Schmalz T, Ludwigs E. Objectifying the functional advantages of prosthetic wrist flexion. J Prosthet Orthot. 2009;21(2):74-8.
- [Background] Deijs M, Bongers RM, Ringeling-van Leusen ND, van der Sluis CK. Flexible and static wrist units in upper limb prosthesis users: functionality scores, user satisfaction and compensatory movements. J Neuroeng Rehabil. 2016 Mar 15;13:26. doi: 10.1186/s12984-016-0130-0. PMID 26979272
- [Background] Resnik L, Borgia M, reliability and validity of outcome measures for upper limb amputation. JPO. 2012;24:192-201
- [Background] Hebert JS, Lewicke J, Williams TR, Vette AH. Normative data for modified Box and Blocks test measuring upper-limb function via motion capture. J Rehabil Res Dev. 2014;51(6):918-32. doi: 10.1682/JRRD.2013.10.0228. PMID 25356979
- [Background] Haverkate L, Smit G, Plettenburg DH. Assessment of body-powered upper limb prostheses by able-bodied subjects, using the Box and Blocks Test and the Nine-Hole Peg Test. Prosthet Orthot Int. 2016 Feb;40(1):109-16. doi: 10.1177/0309364614554030. Epub 2014 Oct 21. PMID 25336050
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Carey SL, Jason Highsmith M, Maitland ME, Dubey RV. Compensatory movements of transradial prosthesis users during common tasks. Clin Biomech (Bristol). 2008 Nov;23(9):1128-35. doi: 10.1016/j.clinbiomech.2008.05.008. PMID 18675497
- [Background] Bouwsema H, van der Sluis CK, Bongers RM. Movement characteristics of upper extremity prostheses during basic goal-directed tasks. Clin Biomech (Bristol). 2010 Jul;25(6):523-9. doi: 10.1016/j.clinbiomech.2010.02.011. Epub 2010 Apr 1. PMID 20362374
- [Background] Loiret I, Paysant J, Martinet N, Andre JM. [Evaluation of amputees]. Ann Readapt Med Phys. 2005 Jul;48(6):307-16. doi: 10.1016/j.annrmp.2005.03.009. Epub 2005 Apr 15. French. PMID 15932782
- [Background] Demers L, Weiss-Lambrou R, Ska B. Development of the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST). Assist Technol. 1996;8(1):3-13. doi: 10.1080/10400435.1996.10132268. PMID 10159726
- [Background] Miller LA, Stubblefield KA, Lipschutz RD, Lock BA, Kuiken TA. Improved myoelectric prosthesis control using targeted reinnervation surgery: a case series. IEEE Trans Neural Syst Rehabil Eng. 2008 Feb;16(1):46-50. doi: 10.1109/TNSRE.2007.911817. PMID 18303805
- [Background] Gouzien A, de Vignemont F, Touillet A, Martinet N, De Graaf J, Jarrasse N, Roby-Brami A. Reachability and the sense of embodiment in amputees using prostheses. Sci Rep. 2017 Jul 10;7(1):4999. doi: 10.1038/s41598-017-05094-6. PMID 28694439